CLINICAL TRIAL: NCT04060745
Title: Glucose Metabolism in Brown Adipose Tissue (BAT) in Young Healthy Men Evaluated by Deuterium Metabolic Imaging (DMI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: MR protocol was not ready for the study. Grant for the study expired.
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Brown fat imaging
Record Dates: First submitted 2019-08-08; First posted 2019-08-19 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2021-05

CONDITIONS: Type2 Diabetes; Obesity; Metabolic Syndrome
Keywords: brown adipose tissue; deuterium metabolic imaging; FDG PET/CT; individualized cooling protocol
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Calorimetry, Indirect

STUDY DESIGN:
Intervention Model Description: Participants will be screened for active brown adipose tissue (BAT) using FDG PET/CT. Only BAT-positive participants will enter the two-phased randomized crossover trial using DMI under cold or thermoneutral conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling (Experimental): Participants will be cooled using an individualized cooling protocol with a water-perfused vest for two hours while resting. Afterwards, participants will drink 75g of D2-glucose dissolved in water and DMI will be performed.
  Interventions: Other: cooling using a water-perfused vest
- Thermoneutrality (Experimental): Participants will rest for one hours. Afterwards, participants will drink 75g of D2-glucose dissolved in water and DMI will be performed.
  Interventions: Other: thermoneutrality

INTERVENTIONS:
Other: cooling using a water-perfused vest — BAT is activated by cold exposure. Each participant will have a shivering threshold test performed before entering the cooling arm. Participants will be gradually cooled (decreasing the temperature in the cooling vest by 0.6C every 15 min. until 3.8C) using a perfused cooling vest until they start to shiver. The temperature in which they start to shiver will be noted. If shivering has not occurred at 3.8C after 15 min. they will stay at the temperature for 45 min. in total or until shivering occurs. Shivering is defined by subjective perception of shivering by the participant in a numeric scale (NRS) where "0" refers to "I'm not shivering" and 10 refers to "I'm shivering a lot" and visual inspection by the investigator. The temperature used in the cooling arm will be set a few degrees above the shivering threshold test or at 3.8C if shivering did not occur.
  During cooling indirect calorimetry and OGTT will be performed and finally the DMI scan will be performed
  Other Names: Indirect calorimetry; oral glucose tollearnce test (OGTT); DMI scan
  Arms: Cooling
Other: thermoneutrality — In the thermoneutrality arm participants will rest in thermoneutrality (22C) for one hour. Before the DMI scan indirect calorimetry will be performed
  Other Names: Indirect calometry; DMI scan
  Arms: Thermoneutrality

SUMMARY:
In this study the investigators wish to evaluate the glucose metabolism in brown adipose tissue (BAT) in young healthy men (aged 18-35). The investigators wish to validate a novel MR modality - Deuterium Metabolic Imaging (DMI), which is a non-radioactive, non-invasive method that allows for spatial as well as metabolic imaging after oral administration of deuterium-labelled glucose. Deuterium is a stable isotope of hydrogen that can be bound to different metabolites, in this case glucose. This method allows for metabolic imaging and production of 2H MR spectra of metabolites downstream from glucose uptake that can be quantified. DMI has not yet been used to evaluate BAT in humans. Currently, FDG PET/CT is the most widely used method for BAT evaluation in humans, but due to the radiation-exposure associated with FDG PET/CT repetitive studies of BAT in healthy subjects are limited. Therefore, new in vivo methods (preferably non-invasive) are warranted.

However, since FDG PET/CT is the most widely used method, the investigators wish to use this modality as reference.

The investigators plan to screen 10-12 subjects with an individualized cooling protocol and FDG PET/CT. Only the BAT positive subjects will be included in the DMI study. In the DMI study, the BAT positive subjects will enter in a randomized two-phased cross-over study. The subjects will have 2 DMI scans performed after ingestion of deuterium-labelled glucose; one after 2h of cooling, another in thermoneutrality. Primary outcome is the differences in glucose metabolites between cooling and thermoneutrality. The investigators hypothesize that during cooling uptake of glucose and its metabolites such as glutamine/glutamate and water may be enhanced. Moreover, glucose metabolism may shift towards anaerobic metabolism with increased lactate production as observed in a previous rodent study by the investigators group.

DETAILED DESCRIPTION:
The prevalence of obesity and type 2 diabetes has increased exponentially over the past decades giving rise to substantial individual as well as health economic costs. Therefore, more research are warranted in the development of new prevention and treatment strategies.

In 2009 findings using 2-deoxy-2-(18F)fluoro-D-glucose positron emission tomography (FDG-PET) verified the presence of metabolically active brown adipose tissue (BAT) in adult humans and since then BAT has been revitalized as a potential target organ in the treatment of obesity and metabolic syndrome. Through increased activity of the sympathetic nervous system (SNS) and the corresponding release of norepinephrine (NE), cold is among the most potent physiological activators of BAT, but other stimulating factors such as natriuretic peptides, BMP8b, COX2, bile acids, thyroid hormones, FGF21 and even bioactive food components are known. Activated BAT increases the energy expenditure via uncoupling (via uncoupling protein 1 - UCP1) of the inner mitochondrial membrane resulting in leak of electrons and heat production at the expense of ATP production (non-shivering thermogenesis) a mechanism evolutionary developed to sustain body temperature. It is known that age, gender, degree of obesity and insulin resistance is associated with BAT activity. Furthermore, activated BAT generally improves glucose tolerance, insulin sensitivity and promotes weight loss in rodent models giving rise to hopes for similar effects in humans. However, deeper insight into in vivo BAT metabolism in humans are still warranted. BAT is anatomically located along the major vessels, surrounding the large organs, the anterior neck, sub-clavicular, axillary and in the inguinal fossa. In this proposed clinical study, the investigators wish to examine the anterior neck and supraclavicular area that are known to comprise the largest BAT depots.

When BAT is activated glucose- as well as free fatty acids uptake are greatly increased compared to non-activated BAT and therefore the most widely used method for in vivo assessment of BAT activity and imaging in humans is currently FDG PET/CT. This well-known imaging modality relies on the radioactive glucose tracer 18FDG to detect tissues with high glucose consumption e.g. activated BAT. The 18FDG signal gives an indication of the distribution of glucose uptake and phosphorylation in the tissue. However, FDG PET imaging does neither provide information on spatial metabolic activity, nor the different metabolites downstream from glucose as FDG is not further metabolized when taken up in the tissue. Moreover, due to the radiation-exposure associated with FDG PET/CT repetitive studies of BAT in healthy subjects are limited.

New in vivo methods (preferably non-invasive) are warranted in order to reveal the true potential of targeting BAT thermogenesis to prevent and/or treat cardio metabolic disorder.

To accommodate this need, Deuterium Metabolic Imaging (DMI) may be a potential tool. DMI is a novel non-radioactive, non-invasive method that allows for spatial as well as metabolic imaging after oral administration of [6,6'- H ]-glucose. Deuterium is a stable isotope of hydrogen that can be bound to different metabolites, in this case glucose. This method allows for metabolic imaging and production of 2H MR spectra of metabolites downstream from glucose uptake that can be quantified. The method has already been applied in studies of the human and rat brain using spectroscopic imaging at 4T and 11.7T respectively, but has never been used to assess glucose metabolism in human BAT.

The acquired spectra from DMI contain peaks of [2H]glucose, [2H]lactate, [2H]-Glx, which contains signals from [4,4´-2H2]glutamate, [4-2H]glutamate, [4´-2H]glutamate, [4,4´-2H2]glutamine, [4´-2H]glutamine and [4´-2H]glutamine and finally [2H]water.

The biochemical pathway of the labelled [2H] is as followed: When [6,6'- 2H2 ]-glucose is taken up in the tissue the [2H] is firstly incorporated into pyruvate to form [3,3-2H]Pyruvate through glycolysis. Under anaerobic circumstances [3,3-2H]Pyruvate is secondly converted to [3,3-2H]lactate catalyzed by lactate dehydrogenase (LDH). [3,3-2H]Pyruvate can also be transported into the mitochondria and be transformed into [2,2-2H]Acetyl-CoA catalyzed by pyruvate dehydrogenase (PDH). When entered into the TCA cycle, the intermediates of [4-2H] or [4,4-2H]Citrate and [4-H] or [4,4-2H]α-ketoglutarate will be produced. The latter may exchange with glutamate to generate [4-H] or [4,4-2H2]glutamate. From the TCA cycle, 2H-labeling may depart and exchange with the protons in water molecules to generate [2H]water.

Prior to this proposed clinical trial, the investigators have recently conducted a rodent study to test the method (data not yet published).

The investigators show that DMI of the interscapular BAT depot in cold-acclimatized rats reveals increases in all [²H]-labelled metabolites after [6,6'-²H₂]-glucose infusion (glucose, glutamine/glutamate, lactate and water) indicating an overall increase in uptake and glucose metabolism with higher glutamine/glutamate and lactate production in cold acclimatized rats compared to thermo-neutral rats. These metabolites potentially originate from an elevated TCA cycle flux and an associated increased anaerobic metabolism in the cold-acclimatized rats. The investigators hereby show that DMI can be used to discriminate between activated and non-activated BAT in rats. These findings are supported by increased mean fat/water threshold in cold-acclimatized rats compared to thermo-neutral rats indicating an increased water content or vascularization. Furthermore, a robust 13-fold increment in the specific thermogenic marker uncoupling protein one (UCP1) mRNA expression was found in BAT biopsy material of cold-acclimatized rats.

These results indicate that DMI of BAT in humans are feasible.

Aim/perspectives To evaluate if DMI can be used to assess and discriminate glucose metabolism in activated and non-activated BAT in humans using a randomized controlled crossover design in healthy young men in order to use this method to determine BAT activity in humans .

The investigators hypothesize that in cold activated BAT glucose metabolism will increase as measured by increase in uptake and metabolism resulting in increase in glucose, glutamate/glutamine and water. Moreover, glucose metabolism may shift from aerobic metabolism towards anaerobic metabolism with increased lactate production in activated BAT as observed in the rodent study.

This non-invasive, non-radioactive method may pave the way for future, repetitive metabolic imaging in humans, which may be an important tool in the development of drugs targeting BAT. Given the relative ease of implementation in a clinical setting and the range of available H-labeled substrates, DMI has the potential to become a widespread MRI modality for metabolic imaging in general.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men (aged 18-35), body mass index (BMI) 18.5-25, weight change ˂ 5% in the last 6 months

Exclusion Criteria:

* acute or chronic disease, regular medication that could influence the cardiovascular or thermoregulatory response, alcohol intake ˃ 21 units/week, claustrophobia, pacemaker or metal devices in the body and smoking.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in glucose metabolism between non-activated and cold-activated BAT | 1-2 weeks
  Changes measured by abundant [2H] labelled glucose signal in non-activated or cold-activated BAT compared to [2H] labelled glucose signal after [2H] labelled glucose ingestion. Delta [2H] labelled glucose signal in the two states will be compared by paired t-test
Changes in glucose metabolism between non-activated and cold-activated BAT | 1-2 weeks
  Changes measured by abundant [2H] labelled lactate signal in non-activated or cold-activated BAT compared to [2H] labelled lactate signal after [2H] labelled glucose ingestion. Delta [2H] labelled lactate signal in the two states will be compared by paired t-test
Changes in glucose metabolism between non-activated and cold-activated BAT | 1-2 weeks
  Changes measured by abundant [2H] labelled glutamate/glutamine signal in non-activated or cold-activated BAT compared to [2H] labelled glutamate/glutamine signal after [2H] labelled glucose ingestion. Delta [2H] labelled glutamate/glutamine signal in the two states will be compared by paired t-test
Changes in glucose metabolism between non-activated and cold-activated BAT | 1-2 weeks
  Changes measured by abundant [2H] labelled water signal in non-activated or cold-activated BAT compared to [2H] labelled water signal after [2H] labelled glucose ingestion. Delta [2H] labelled water signal in the two states will be compared by paired t-test

SECONDARY OUTCOMES:
BAT DMI measurements compared to plasma NMR measurements | 1-2 weeks
  Correlations between [2H] labelled glucose in plasma versus BAT measured by [2H] signal change
BAT DMI measurements compared to plasma NMR measurements | 1-2 weeks
  Correlations between [2H] labelled lactate in plasma versus BAT measured by [2H] signal change
BAT DMI measurements compared to plasma NMR measurements | 1-2 weeks
  Correlations between [2H] labelled glutamate/glutamine in plasma versus BAT measured by [2H] signal change
BAT DMI measurements compared to plasma NMR measurements | 1-2 weeks
  Correlations between [2H] labelled water in plasma versus BAT measured by [2H] signal change
Changes in fat/water thresholds in BAT in cold versus thermoneutral conditions | 1-2 weeks
  Changes in fat/water thresholds in BAT measured by Dixon MRI, fat/fat+water signal x 100%
Changes in metabolic profiles in cold versus thermoneutral conditions | 3-4 weeks
  Changes in plasma glucose in cold versus thermoneutral conditions, units: mmol/L
Changes in metabolic profiles in cold versus thermoneutral conditions | 3-4 weeks
  Changes in plasma fatty acids in cold versus thermoneutral conditions, units mmol/L
Changes in metabolic profiles in cold versus thermoneutral conditions | 3-4 weeks
  Changes in plasma insulin levels in cold versus thermoneutral conditions, units pmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided